## Utility of an Animated Bowel Biofeedback Training Routine to Improve Bowel Function in Individuals With SCI

NCT02406859

March 10, 2013

## **Statistical Analysis Plan**

For the continuous dependent, independent and demographic variables, descriptive statistics will be performed and expressed as group mean ± SD, with 95% confidence intervals and ranges. To examine the effect of the training on manometric and subjective parameters (groups: stratified by level of injury and completeness) analysis of variance (ANOVA) with repeated measures on visit (Pre, Post) will be performed. In the event of non-normal distribution of study outcomes, non-parametric ranking statistics will be applied as appropriate. An a priori level of significance will be set at P≤0.05. IBM SPSS Statistics version 22 will be used for all analyses.